CLINICAL TRIAL: NCT06187402
Title: A Phase I/II, First-in-Human (FIH), Open-Label, Multiple Centre Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy of LM-24C5 in Patients With Advanced Solid Tumors
Brief Title: A Study of LM-24C5 For Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LaNova Medicines Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LM24C5-01-101
Record Dates: First submitted 2023-12-04; First posted 2024-01-02 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LM-24C5 Dose Escalation (Experimental)
  Interventions: Drug: LM-24C5
- LM-24C5 Dose Expansion (Experimental)
  Interventions: Drug: LM-24C5

INTERVENTIONS:
Drug: LM-24C5 — Administered intravenously

SUMMARY:
To assess the safety and tolerability, obtain the recommended phase 2 dose (RP2D)/optimal biologic dose (OBD) and/or Maximum Tolerated Dose (MTD) for LM-24C5 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are fully informed of the purpose, nature, method and possible adverse reactions of the study, and are willing to participate in the study and sign the informed consent form (ICF) prior to any study related procedures.
2. Aged ≥18 years old when sign the ICF, male or female.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, and no deterioration within 2 weeks prior to the first dose.
4. Life expectancy ≥ 3 months.
5. Subjects must have histological or cytological confirmation of recurrent or refractory advanced solid tumors, and have progressed on standard therapy, or are intolerable for available standard therapy, or there is no available standard therapy.
6. Formalin-fixed paraffin-embedded (FFPE) tumor tissue samples meet the minimum requirements.
7. At least one measurable lesion according to RECIST v1.1.
8. Subjects must show appropriate organ and marrow function in laboratory examinations within 7 days prior to the first dose.
9. Subjects who are able to communicate well with investigators and understand and adhere to the requirements of this study.

Exclusion Criteria:

1. Participate in any other clinical trial within 28 days prior to 1st dosing of LM-24C5.
2. Any prior treatments towards the investigational target.
3. Subjects with anti-tumor treatment within 21 days prior to 1st dosing of LM-24C5, including radiotherapy, chemotherapy, biotherapy, endocrine therapy and immunotherapy, etc. the following treatments have different time limits.
4. Any adverse event from prior anti-tumor therapy has not yet recovered to≤ grade 1 of CTCAE v5.0.
5. Subjects with uncontrolled pain.
6. Subjects with known central nervous system (CNS) or meningeal metastasis.
7. Subjects who have uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
8. Subjects who experienced grade 3 or higher hypersensitivity to the treatment that contains any monoclonal antibody.
9. Subjects who take systemic corticosteroids (> 10 mg daily prednisone equivalents) or other systemic immunosuppressive medications within 2 weeks prior to the first dosing of LM-24C5.
10. Subjects with the known history of autoimmune disease.
11. Subjects with the history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
12. Use of any live attenuated vaccines within 28 days prior to 1st dosing of LM-24C5.
13. Subjects who are taking therapeutic doses of anticoagulants such as heparin or vitamin K antagonists for presence of active thromboembolic disease.
14. Subjects who received major surgery or interventional treatment within 28 days prior to 1st dosing of LM-24C5.
15. Subjects who have severe cardiovascular disease.
16. Subjects who have uncontrolled or severe illness, including but not limited to ongoing or active infection
17. Subjects who have a history of immunodeficiency disease, including other acquired or congenital immunodeficiency diseases, or organ transplantation, or allogeneic bone marrow transplantation, or autologous hematopoietic stem cell transplantation.
18. HIV infection, active infection including tuberculosis, HBV and HCV infection, with the exception:
19. Subjects who have other active malignancies which are likely to require the treatment.
20. Child-bearing potential female who have positive results in pregnancy test or are lactating.
21. Subjects who have psychiatric illness or disorders that may preclude study compliance.
22. Subject who is judged as not eligible to participate in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 60 weeks
  Phase 1
Incidence of dose-limiting toxicity (DLT) | 60 weeks
  Phase 1
Incidence of serious adverse event (SAE) | 60 weeks
  Phase 1
Ear Temperature | 60 weeks
  Phase 1
Pulse in BPM(Beat per Minute) | 60 weeks
  Phase 1
Blood Pressure in mmHg (Both Systolic and Diastolic blood pressure) | 60 weeks
  Phase 1
Number of participants with abnormal Hematology test results | 60 weeks
  Phase 1
Number of participants with abnormal Urinalysis test results | 60 weeks
  Phase 1
Number of participants with abnormal Blood Biochemistry test results | 60 weeks
  Phase 1
Number of participants with abnormal Coagulation test results in PT(Prothrombin time), APTT(Activated partial thromboplastin time), FIB(Fibrinogen), TT(Thrombin time) and INR(International normalized ratio). | 60 weeks
  Phase 1
Echocardiography- LVEF(Left Ventricular Ejection Fraction) in percentage | 60 weeks
  Phase 1
12-lead electrocardiogram (ECG) in RR, PR, QRS, QT, QTcF etc. | 60 weeks
  Phase 1
ECOG(Eastern Cooperative Oncology Group) score | 60 weeks
  Phase 1
Overall Response Rate (ORR) | 36 weeks
  Phase 2

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameter: Maximum Observed Concentration (Cmax) | 96 weeks
  Phase 1 and 2
PK Parameter:Time of Maximum Observed Concentration (Tmax) | 96 weeks
  Phase 1 and 2
PK Parameter: Area Under the Concentration-time Curve(AUC) | 96 weeks
  Phase 1 and 2
PK Parameter: Steady State Maximum Concentration(Cmax,ss) | 96 weeks
  Phase 1 and 2
PK Parameter: Steady State Minimum Concentration(Cmin,ss) | 96 weeks
  Phase 1 and 2
PK Parameter: Systemic Clearance at Steady State (CLss) | 96 weeks
  Phase 1 and 2
PK Parameter: Accumulation Ratio (Rac) | 96 weeks
  Phase 1 and 2
PK Parameter: Elimination Half-life (t1/2) | 96 weeks
  Phase 1 and 2
PK Parameter: Volume of Distribution at Steady-State (Vss) | 96 weeks
  Phase 1 and 2
PK Parameter: Degree of Fluctuation (DF) | 96 weeks
  Phase 1 and 2
Immunogenicity of LM-24C5 | 96 weeks
  Phase 1 and 2; Anti-Drug antibody and Nab (if necessary) will be tested.
Duration of Response (DOR) in Month | 96 weeks
  Phase 1 and 2
Disease control rate (DCR) in percentage | 96 weeks
  Phase 1 and 2
progression-free survival (PFS) in Month | 96 weeks
  Phase 1 and 2
Overall survival (OS) in Month | 60 weeks
  Phase 1
Changes of target lesions from baseline in Millimeter. | 96 weeks
  Phase 1 and 2
Safety: AE/SAE (Number of participants with treatment-related adverse events as assessed by CTCAE v5.0) | 36 weeks
  Phase 2
Ear Temperature | 36 weeks
  Phase 2
Pulse in BPM (Beat per Minute) | 36 weeks
  Phase 2
Blood Pressure in mmHg (Both Systolic and Diastolic blood pressure) | 36 weeks
  Phase 2
Number of participants with abnormal Hematology test results | 36 weeks
  Phase 2
Number of participants with abnormal Urinalysis test results | 36 weeks
  Phase 2
Number of participants with abnormal Blood Biochemistry test results | 36 weeks
  Phase 2
Number of participants with abnormal Coagulation test results in PT(Prothrombin time), APTT(Activated partial thromboplastin time), FIB(Fibrinogen), TT(Thrombin time) and INR(International normalized ratio). | 36 weeks
  Phase 2
12-lead electrocardiogram (ECG) in RR, PR, QRS, QT, QTcF etc. | 36 weeks
  Phase 2
ECOG(Eastern Cooperative Oncology Group) score | 36 weeks
  Phase 2

OTHER OUTCOMES:
Relationship between the biomarkers and the anti-tumor activity | 96 weeks
  Phase 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Terry Pang, Study Director — LaNova
Locations (6):
- United States (6):
  - University of Southern California (USC) - Norris Comprehensive Cancer Center, Los Angeles, California
  - Ocala Oncology, Ocala, Florida
  - Indiana University Melvan and Bren Simon Cancer Center, Indianapolis, Indiana
  - The Christ Hospital, Cincinnati, Ohio
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - Virginia Cancer Specialists, P.C., Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No